CLINICAL TRIAL: NCT05347654
Title: Evaluation of a Management Strategy for Second-degree Fibrinous Burns Integrating a Poly-absorbent Dressing: a Prospective, Controlled, Open, Randomized Multicentre Study
Brief Title: Evaluation of a Management Strategy for Second-degree Fibrinous Burns Integrating a Poly-absorbent Dressing
Acronym: HYDRA-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0076
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Burns Degree Second
Keywords: Burns Degree Second; detersion,; poly-absorbent dressing; wound healing; skin graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard strategy (Active Comparator): Local treatment with silver sulphadiazine and tulle from day 0 to day 8. From the 9t h day and until healing, the dressings are made with tulle, every 48 hours.
  Interventions: Other: Local treatment with silver sulphadiazine only
- Strategy incorporating a poly-absorbent dressing (Experimental): Local treatment of silver sulphadiazine with tulle from day 0 to day 4, then with URGOCLEAN® dressing every 48h from day 5 to day 8. From the 9th day and until healing, the dressings are made with tulle, every 48 hours.
  Interventions: Other: Local treatment with silver sulphadiazine followed by URGOCLEAN® dressing

INTERVENTIONS:
Other: Local treatment with silver sulphadiazine only — Local treatment with silver sulphadiazine and tulle from day 0 to day 8 (included). From the 9th day and until healing, the dressings are made with tulle, every 48 hours.
  Arms: Standard strategy
Other: Local treatment with silver sulphadiazine followed by URGOCLEAN® dressing — Local treatment of silver sulphadiazine with tulle from day 0 to day 4, then with URGOCLEAN® dressing every 48h from day 5 to day 8. From the 9th day and until healing, the dressings are made with tulle, every 48 hours.
  Arms: Strategy incorporating a poly-absorbent dressing

SUMMARY:
The management of the local treatment of second-degree burns has an influence on the healing time and thus on the quality of the healing process. Fibrin detersion optimizes epidermization and may reduce the need for skin grafting for moderate fibrinous burns. Optimal treatment at this stage is therefore crucial. Since 1968, silver sulphadiazine ointment dressings have been used in the management of burns to minimize the risk of infection. A recent review of the literature suggests that the use of alternative dressings to silver sulphadiazine ointment, from day 3/4, would have a benefit on wound healing, but highlights the insufficient level of evidence in current studies. This probably explains why the prolonged use of silver sulphadiazine dressings remains the rule in the majority of French centres. In the burns department of Hopital Edouard Herriot, PLASTENAN® ointment was used as a relay to silver sulphadiazine after one week of care to promote the detersion of second-degree fibrinous burns. Following the end of its commercialization in 2014, our nursing team wondered whether an ointment or an equivalent dressing was available. A clinical study on URGOCLEAN® dressing was conducted by another team from our university hospital on the detersion of vascular wounds. Given its positive results,the investigator tested its effectiveness on fibrinous burns. A cohort of 70 patients (2014-2018) was thus set up by our nursing team: this dressing used in fibrinous burns showed a low use of skin grafts (2/70), a median healing time of 20 days and an improvement in the quality of the scar. In 2013, a systematic review by the Cochrane compared seven types of dressings for the treatment of superficial and intermediate burns, but the URGOCLEAN® dressing, marketed in 2013, was not included. Considering these findings, the investigator would like to set up a randomized trial to evaluate a strategy integrating the URGOCLEAN® dressing in the management of second-degree fibrinous burns.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* 2nd degree burn with : Affected body surface between 0.25 et 10% Fibrinous surface between 9 and 156 centimeter/meter square (major axis between 3 and 16 centimeter, minor axis of 3 centimeter minimum) One or more non-contiguous fibrinous surfaces
* Exudative wet fibrin
* Patient treated with silver sulphadiazine between Day 0 and Day 4
* Patient affiliated to a social security scheme
* Patient who signed a written consent to participate in the study

Exclusion Criteria:

* Facial burn
* Known diabetic patient
* Patient with severe venous and / or arterial insufficiency (obliterating arteriopathy of the lower limbs stage III and IV)
* Allergy to one of the components of the URGOCLEAN® dressing (polyacrylate fibers, carboxymethylcellulose, paraffin oil, petroleum jelly)
* Person under guardianship or curators
* Patient deprived of liberty
* Patient for whom silver sulphadiazine is contraindicated (last trimester of pregnancy, lactating woman, allergy to sulfa drugs)
* Patient treated with pre-impregnated interfaces (URGOTUL SAG®, IALUSET+® compresses,..) during initial care between Day 0 and Day 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Number of patients with a skin graft performed before D21 | At day 21
  The number of patients with a skin graft performed before D21 will be calculated. In case the graft is indicated but the patient refuses it, he will be counted as having had a graft.

SECONDARY OUTCOMES:
Quality of the scar according to health professional | at 1 month, at 3 months, at 6 months, at 12 months
  The quality of the scar according to the professional will be assessed using the total POSAS (Patient and Observer Scar Assessment Scale ) score. Score from 7 (best score) to 70 (worst score)
Scar quality according to patient | at 1 month, at 3 months, at 6 months, at 12 months
  The quality of the scar according to the patient will be assessed using the total POSAS (patient) score. Score from 7 (best score) to 70 (worst score)
Complete healing for non-grafted patients | at day 21
  Complete healing for non-grafted patients assessed by the number of patients with epidermization defined by total wound coverage with pink epithelium and dressing discontinuation
Complete healing | at 3 months, at 6 months, at 12 months
  The number of patients for whom scar healing is observed will be calculated. Scar healing is defined by: dressing discontinuation, and scar maturation (cessation of compression), and clinical follow-up discontinuation.
Dressing tolerance | at Day 5, Day 6, Day 7, Day 8
  Any dressing discontinuation related to adverse events, and all tolerance events observed during the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, Rhone, France